CLINICAL TRIAL: NCT01143935
Title: Estimation of Standard Liver Volume in the Indian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr Gaurav Nitin Chaubal, AIIMS
Other Study IDs: liver volume estimation
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-01

CONDITIONS: Liver
Keywords: Liver volume estimation; Indian population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Live patients: All patients undergoing CT scans of the abdomen for non hepatobiliary conditions
- Autopsy cases: All autopsy cases with no liver disease or trauma.

SUMMARY:
Estimation of liver volume is important for live donor liver transplant as well as extended liver resections. Computed tomography (CT) volumetry which is currently a gold standard for liver volumetry , is a time consuming process. A quicker method to estimate liver volume is essential. The aim of the present study is to try and formulate an equation based on patients height, weight etc to estimate liver volume.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing CT scans

* Autopsy cases

Exclusion Criteria:

* Patients with hepatobiliary disorders Autopsy cases with liver disease or trauma

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing CT scans for non hepatobiliary conditions. Autopsy cases in whom there is no liver disease or trauma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tushar K Chattopadhyaya, MS Surgery, Study Chair — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India